CLINICAL TRIAL: NCT05865262
Title: Analysis of Ventricular Repolarization by QT Measurement in Transgender People Treated With Hormone Therapy
Brief Title: Protocol TRANS and QT Repolarization
Acronym: QTrans
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: APHP (Other)
Responsible Party: Principal Investigator, Virginie GROUTHIER, Principal Investigator Medical doctor, University Hospital, Bordeaux
Other Study IDs: 2021.11.16_Grouthier
Record Dates: First submitted 2023-04-26; First posted 2023-05-18 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Transgender Individuals; QTc Interval
Keywords: Transgender; QTc; testoterone; estradiol; ventricular repolarization
MeSH Terms: interventions — Electrocardiography; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- treated transgender people: Transgender individuals consulting at the Endocrinology department of the Haut-Leveque hospital in Pessac (France), whether they are (one unique visit) or not (2 visits) already on GAHT (feminizing hormone treatment in transgender women and masculinizing treatment in transgender men, respectively). Men and women not already on GAHT will have two visits in total, one inclusion visit before GAHT start and one at least after one month of GAHT (and maximum within 2 years of start). Transgender individuals already on GAHT will have one unique inclusion visit without any planned follow-up visit.
  Interventions: Diagnostic Test: ECG; Diagnostic Test: blood test (assessing ionic and hormonal circulating levels)

INTERVENTIONS:
Diagnostic Test: ECG — A triplicate ECG and a blood test will be done during a medical consultation as part of the usual endocrinology follow-up. Included individuals seen prior to initiation of GAHT, will be assessed a second time (at least one month after GAHT start) with a triplicate ECG and a blood test similar to inclusion visit. Included individuals already on GAHT will be seen only once at the inclusion visit.
  Triplicates of 10seconds 12-lead digitized electrocardiogram will be recorded after few minutes of rest in the supine position. Electrocardiograms will be acquired with Mindray ECG BeneHeart R12. For each subject, RR, PR, QRS and QT interval durations will be assessed with a semiautomatic approach using the median representative beats (overlap method) generated from 10seconds ECG with a good quality (CalECG v3.7; AMPS, LLC). The QT interval will be measured and corrected for heart rate by Fridericia's formula.
Diagnostic Test: blood test (assessing ionic and hormonal circulating levels) — Blood samples for the determination of serum concentrations of estradiol, progesterone, testosterone, FSH, and LH will be collected on the same day as the ECG, in a dry tube and further assayed in the immunology laboratory of Bordeaux University Hospital (France). Estradiol, progesterone, FSH, and LH plasma concentrations will be assayed by immunochemiluminescence (Architect i2000SR; Roche Diagnostics), and testosterone levels by liquid chromatography mass spectrometry. Kalemia and calcemia will be collected in a BD Vacutainer tube with heparin lithium and separator, further assayed at the biochemistry laboratory of Bordeaux University Hospital by indirect potentiometric measurement (Architect c16000) and Arsenazo III SRM 956 colorimetrie (Architect c16000).

SUMMARY:
The consequence of hormone-based treatment on cardiac electrophysiology in transgender individuals is poorly explored. We will investigate the effects of gender affirming hormone treatments on ventricular repolarization (ie. QTc, QT corrected for heart rate duration) in a prospective cohort of transgender individuals before and after feminizing and masculinizing treatments, and transversally in transgender individuals on gender affirming hormone treatments. This monocentric cohort will be included in the Endocrinology department of the Haut-Leveque Hospital in Pessac (France).

DETAILED DESCRIPTION:
An essential step in the care of gender dysphoria is gender-affirming hormone therapy (GAHT) combining an anti-androgen and estrogen therapy in transgender women (formerly male to female) or androgen therapy in transgender men (female to male). Several studies have shown a detrimental effect of GAHT on cardiovascular risk factors and therefore, the European Society of Endocrinology recommend an enhanced monitoring of cardiovascular risk factors in transgender population. Data on the risk of cardiac arrhythmias in transgender population are lacking, particularly on ventricular repolarization and QTc.

Indeed, sex steroid hormones and gonadotropins are known to alter the cardiac electrophysiology, as shown in various animal and human studies. From puberty to menopause, the QTc is generally longer in women than in men, translating into a higher risk of Torsade de Pointes (a peculiar form of ventricular arrhythmia) in women versus men. Recent publications have well illustrated the shortening of QTc in women in situation of biological hyperandrogenism and; QTc lengthening in hypogonadal men which was reversed by restoration of physiological eugonadal testosterone levels. Gonadotrophin's levels were positively correlated with QTc. To date, no study has focused on changes in cardiac repolarization in the transgender population and particularly on the effects of GAHT.

The aim of this study is to evaluate the impact of feminizing and masculinizing hormone treatments (GAHT) on ventricular repolarization (i.e QTc) in transgender individuals, followed at the Endocrinology department of the Haut-Leveque hospital in Pessac.

We aim to enroll consecutively (monocentric cohort) transgender individuals (on and before treatment) consulting to the endocrinology department for their usual standard of care follow-up until we include 15 transgender men and 15 transgender women with 2 QTc assessments available, one before and the other after initiation of GAHT (triplicates of 10 sec ECGs, Fridericia's heart rate correction for each time-point). This effective (n=15/group) have ≥85% power to detect a difference in QTcF≥10msec between the ECG before and after initiation of GAHT with a paired t-test (α: 0.05; standard deviation of QTc in each subgroup: 12msec; expected QTcF mean: 410msec and 400msec in women and men before GAHT, respectively, intra-individual correlation: 0.5).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with gender dysphoria consulting as part of the usual standard of care follow-up in endocrinology for instauration of the follow-up of GAHT

Exclusion Criteria:

* <18 years old
* patients under protective measures or deprived of liberty (under guardianship, curatorship, safeguard of justice, incarcerated)
* history of congenital long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with gender dysphoria consulting as part of the usual standard of care follow-up in endocrinology for instauration or follow-up of GAHT
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
To assess the impact of GAHT on QTc duration in transgender individuals before and after starting therapy | assessments at inclusion and during follow-up visit in endocrinology department (minimum 1 month and max 2 years after treatment started)
  Difference in QTc duration before and after initiation of GAHT

SECONDARY OUTCOMES:
To assess the difference in PR, QRS, RR, QTc duration between men and women prior to GAHT, and transmen and transwomen already on GAHT. | assessments at inclusion and during follow-up visit in endocrinology department (minimum 1 month and max 2 years after treatment started)
  Difference in PR, QRS, RR, QT, QTc duration on digital ECG at initial inclusion visit between men and women prior to GAHT, and transmen and transwomen already on GAHT
To assess the impact of gender-affirming hormone treatment on PR, QRS, RR duration in transgender individuals before and after starting GAHT | assessments at inclusion and during follow-up visit in endocrinology department (minimum 1 month and max 2 years after treatment started)
  Difference in PR, QRS, RR duration before and after initiation of GAHT.
To assess the association between the hormonal and ionic levels with PR, QRS, RR, QTc duration in transgender individuals before and on GAHT. | assessments at inclusion and during follow-up visit in endocrinology department (minimum 1 month and max 2 years after treatment started)
  Correlation (univariate and multivariate, including mixed effects models) between PR, QRS, RR, QTc duration and hormonal (progesterone, testosterone, FSH, LH, estradiol) and ionic (potassium, calcium) circulating levels

CONTACTS AND LOCATIONS:
Overall Officials: Joe-Elie Salem, Pr, Study Chair — Groupe Hospitalier Pitie-Salpetriere
Locations (1):
- University Hospital Bordeaux, France, Pessac, France